CLINICAL TRIAL: NCT05555732
Title: A Randomized Phase 3 Study of Datopotamab Deruxtecan (Dato-DXd) and Pembrolizumab With or Without Platinum Chemotherapy in Subjects With No Prior Therapy for Advanced or Metastatic PD-L1 TPS <50% Non-squamous Non-small Cell Lung Cancer Without Actionable Genomic Alterations (TROPION-Lung07)
Brief Title: Datopotamab Deruxtecan (Dato-DXd) and Pembrolizumab With or Without Platinum Chemotherapy in 1L Non-Small Cell Lung Cancer (TROPION-Lung07)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: AstraZeneca (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS1062-A-U303; 2022-500802-16-00 (Other: EU CT Number); MK3475-C73 (Other: Merck); jRCT Number (Registry Identifier: jRCT2061220066)
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Non Small Cell Lung Cancer
Keywords: Metastatic Non Small Cell Lung Cancer; Advanced Non Small Cell Lung Cancer; Datopotamab Deruxtecan (Dato-DXd); Pembrolizumab; Pemetrexed; Tropion-Lung07
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Pemetrexed; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dato-DXd + Pembrolizumab + Platinum Chemotherapy (Experimental): Participants will be randomized to receive 6.0mg/kg Dato-DXd plus 200 mg pembrolizumab plus platinum chemotherapy (cisplatin 75 mg/m^2 or carboplatin area under the curve [AUC) 5]).
  Interventions: Drug: Datopotamab Deruxtecan; Drug: Pembrolizumab; Drug: Carboplatin; Drug: Cisplatin
- Dato-DXd + Pembrolizumab (Experimental): Participants will be randomized to receive 6.0mg/kg Dato-DXd plus 200 mg pembrolizumab.
  Interventions: Drug: Datopotamab Deruxtecan; Drug: Pembrolizumab
- Pembrolizumab + Pemetrexed + Platinum Chemotherapy (Active Comparator): Participants will be randomized to receive 200 mg pembrolizumab plus 500 mg/m^2 pemetrexed plus platinum chemotherapy (cisplatin 75 mg/m^2 or carboplatin area under the curve [AUC) 5]).
  Interventions: Drug: Pembrolizumab; Drug: Pemetrexed; Drug: Carboplatin; Drug: Cisplatin

INTERVENTIONS:
Drug: Datopotamab Deruxtecan — Dato-DXd will be administered as an intravenous (IV) infusion every 3 weeks on Day 1 of each 21-day cycle.
  Other Names: Dato-DXd
  Arms: Dato-DXd + Pembrolizumab; Dato-DXd + Pembrolizumab + Platinum Chemotherapy
Drug: Pembrolizumab — Pembrolizumab will be administered as an intravenous (IV) infusion every 3 weeks on Day 1 of each 21-day cycle.
  Other Names: KEYTRUDA®
Drug: Pemetrexed — Pemetrexed will be administered as an intravenous (IV) infusion every 3 weeks on Day 1 of each 21-day cycle.
  Other Names: Alimta; Pemfexy
  Arms: Pembrolizumab + Pemetrexed + Platinum Chemotherapy
Drug: Carboplatin — Carboplatin will be administered an intravenous (IV) infusion every 3 weeks on Day 1 of each 21-day cycle for up to 4 cycles.
  Arms: Dato-DXd + Pembrolizumab + Platinum Chemotherapy; Pembrolizumab + Pemetrexed + Platinum Chemotherapy
Drug: Cisplatin — Cisplatin will be administered an intravenous (IV) infusion every 3 weeks on Day 1 of each 21-day cycle for up to 4 cycles.
  Arms: Dato-DXd + Pembrolizumab + Platinum Chemotherapy; Pembrolizumab + Pemetrexed + Platinum Chemotherapy

SUMMARY:
This study is designed to assess the efficacy and safety of datopotamab deruxtecan (Dato-DXd) in combination with pembrolizumab versus pembrolizumab in combination with pemetrexed and platinum chemotherapy in participants with no prior therapy for advanced or metastatic non-squamous non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
The primary objectives of the study are Progression Free Survival (PFS) and Overall Survival (OS) as first line therapy in participants with programmed death-ligand 1 (PD-L1) TPS <50% and advanced or metastatic NSCLC without actionable genomic alternations.

Eligible participants will be randomized in a 1:1:1 ratio to a) Dato-DXd plus pembrolizumab plus platinum; b) Dato-DXd plus pembrolizumab; or c) pembrolizumab plus pemetrexed plus platinum. Platinum therapy will be either carboplatin or cisplatin at investigator discretion. The study will be divided into three periods: Screening Period (including tissue screening), Treatment Period, and Follow-up Period.

ELIGIBILITY:
Key Inclusion Criteria:

1. Sign and date the Main ICF, prior to the start of any study- specific qualification procedures. Is willing and able to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures, and study restrictions.
2. Adults ≥18 at the time the Main ICF is signed. (Follow local regulatory requirements if the legal age of adult voluntary consent for study participation is >18 years old).
3. Has tumor with PD-L1 TPS <50% as determined by PD-L1 IHC 22C3 pharmDx assay by central testing (minimum of six slides). PD-L1 expression results available at the same central laboratory from screening for the purpose of entry into another Dato-DXd study may be used for tissue screening purposes in this study as long as the subject has not been randomized/enrolled in the other study.
4. Has provided a formalin-fixed tumor tissue sample (minimum of 4 × 4-micron sections or block equivalent) for the measurement of TROP2 protein expression and for the assessment of other exploratory biomarkers. This tissue requirement is in addition to the tissue required for PD-L1 testing for tissue screening purposes. If a documented law or regulation prohibits (or does not approve) sample collection, then such sample will not be collected, and the subject is still eligible for the study.
5. Has not been treated with systemic anticancer therapy for advanced or metastatic non-squamous NSCLC. Subjects who received adjuvant or neoadjuvant therapy other than those listed in the exclusion criteria are eligible if the adjuvant/ neoadjuvant therapy was completed at least 6 months prior to the diagnosis of advanced/metastatic disease and should not have progressed on or within the 6 months of completion.
6. Has measurable disease based on local imaging assessment using RECIST v1.1; radiographic tumor assessment must be performed within 28 days before randomization.

Key Exclusion Criteria:

1. Has received prior systemic treatment for advanced/metastatic NSCLC.
2. Has received prior treatment with any of the following, including in the adjuvant/neoadjuvant setting (for NSCLC):

   1. Any agent, including an ADC, containing a chemotherapeutic agent targeting topoisomerase I
   2. TROP2-targeted therapy
   3. Any anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX40, CD137)
   4. Any other ICIs Subjects who received adjuvant or neoadjuvant therapy OTHER than those listed above are eligible if the adjuvant/neoadjuvant therapy was completed at least 6 months prior to the diagnosis of advanced or metastatic disease.
3. Has received a live vaccine within 30 days prior to the first dose of study treatment.

   Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed. For any subject receiving an approved severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) vaccine, please follow the vaccine label and/or local guidance. The vaccine manufacturer and the date of administration should be recorded on the electronic case report form (Concomitant Medications page), as should any AEs relating to the vaccine (including hypersensitivity or allergies). Note: Any licensed SARS-CoV2 vaccine (including those authorized for emergency use) in a particular country is allowed in the study as long as the vaccine is an mRNA vaccine, replication-incompetent adenoviral vaccine, or inactivated vaccine. Such vaccines will be treated just as any other concomitant therapy.

   Investigational vaccines (ie, those not licensed or authorized for emergency use) are not allowed.
4. Has spinal cord compression or clinically active untreated CNS metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are radiologically stable (ie, without evidence of progression) for at least 2 weeks by repeat imaging (Note: Repeat imaging should be performed during study screening), clinically stable, and without requirement of steroid treatment for at least 7 days before the first dose of study drug. Note: A contrasted computed tomography (CT) scan or magnetic resonance imaging (MRI) scan of the brain at baseline (MRI with contrast preferred) is required for all subjects. For those subjects in whom CNS metastases are first discovered at the time of screening, the treating investigator must delay of study treatment to document stability of CNS metastases with repeat imaging at least 2 weeks later (in which case, repeat of all screening activity may be required).
5. Has uncontrolled or significant cardiovascular disease not controlled by maximal medical therapy, including:

   1. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) interval >470 msec regardless of sex (based on the 12-lead electrocardiogram [ECG] performed at screening).
   2. Myocardial infarction within 6 months prior to Cycle 1 Day 1.
   3. History of a serious cardiac arrhythmia requiring treatment
   4. Uncontrolled angina pectoris within 6 months prior to Cycle 1 Day 1.
   5. Left ventricular ejection fraction (LVEF) <50% by echocardiogram (ECHO) or multigated acquisition (MUGA) scan within 28 days before randomization.
   6. New York Heart Association (NYHA) Class II-IV congestive heart failure (CHF) at screening. Subjects with a history of Class II to IV CHF prior to screening, must have returned to Class I CHF and have LVEF ≥50% (by either an ECHO or MUGA scan within 28 days before randomization) in order to be eligible.
   7. Uncontrolled hypertension (resting systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg within 28 days before randomization that is not resolved despite maximal medical therapy).
6. Clinically severe pulmonary compromise as judged by the investigator resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (eg, pulmonary emboli diagnosed within 3 months of Cycle 1 Day 1, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, pleural effusion, etc) or any autoimmune, connective tissue or inflammatory disorders with pulmonary involvement (eg, rheumatoid arthritis, Sjögren's syndrome, sarcoidosis, etc), or prior complete pneumonectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1170 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival Based on Blinded Independent Central Review in Participants With Advanced or Metastatic Non Small Cell Lung Cancer (NSCLC) | From randomization until disease progression or death (whichever occurs first), up to approximately 29 months
  Progression-free Survival (PFS) is defined as the time from randomization to the first documented radiographic disease progression or death due to any cause, whichever occurs first, assessed by blinded independent central review (BICR) per Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1.
Overall Survival in Participants in Participants With Advanced or Metastatic Non Small Cell Lung Cancer (NSCLC) | From randomization until disease progression or death (whichever occurs first), up to approximately 57 months
  Overall Survival (OS) is defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate by Blinded Independent Central Review in Participants With Advanced or Metastatic Non Small Cell Lung Cancer (NSCLC) | From randomization until disease progression or death (whichever occurs first), up to approximately 29 months
  Objective Response Rate (ORR) is defined as the proportion of participants who achieved a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR), assessed by BICR per RECIST Version 1.1.
Progression-free Survival by Investigator in Participants With Advanced or Metastatic Non Small Cell Lung Cancer (NSCLC) | From randomization until disease progression or death (whichever occurs first), up to approximately 29 months
  Progression-free Survival (PFS) is defined as the time from randomization to the first documented radiographic disease progression or death due to any cause, whichever occurs first, assessed by the Investigator per RECIST Version 1.1.
Objective Response Rate by Investigator in Participants With Advanced or Metastatic Non Small Cell Lung Cancer (NSCLC) | From randomization until disease progression or death (whichever occurs first), up to approximately 29 months
  Objective Response Rate (ORR) is defined as the proportion of participants who achieved a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR), assessed by the Investigator per RECIST Version 1.1.
Duration of Response by BICR and Investigator in Participants With Advanced or Metastatic Non Small Cell Lung Cancer (NSCLC) | From date of first objective response (CR or PR) to date of first radiographic disease progression or death due to any cause (whichever occurs first), up to approximately 29 months
  Duration of Response (DoR) is defined as the time from the date of the first documentation of objective response (confirmed CR or confirmed PR) to the date of the first radiographic disease progression or death due to any cause, whichever occurs first, assessed by BICR and by the Investigator per RECIST Version 1.1.
Time to Response by BICR and Investigator in Participants With Advanced or Metastatic Non Small Cell Lung Cancer (NSCLC) | From randomization to date of first objective response (CR or PR), up to approximately 29 months
  Time to Response (TTR) is defined as the time from randomization to the date of the first documentation of objective response (confirmed CR or confirmed PR) in responding participants, assessed by BICR and by the Investigator per RECIST Version 1.1.
Disease Control Rate by BICR and Investigator in Participants With Advanced or Metastatic Non Small Cell Lung Cancer (NSCLC) | From randomization until disease progression or death (whichever occurs first), up to approximately 29 months
  Disease Control Rate (DCR) is defined as the proportion of participants who achieved a BOR of confirmed CR, confirmed PR, or stable disease (SD), assessed by BICR and by the Investigator per RECIST Version 1.1.
Progression-free Survival 2 in Participants With Advanced or Metastatic Non Small Cell Lung Cancer (NSCLC) | From randomization until disease progression or death (whichever occurs first), up to approximately 57 months
  Progression-free Survival 2 (PFS2) is defined as the time from randomization to the first documented radiographic disease progression or death due to any cause, whichever occurs first, assessed by local standard clinical practice
Time to Deterioration in Participants With Advanced or Metastatic Non Small Cell Lung Cancer (NSCLC) | From randomization until disease progression or death (whichever occurs first), up to approximately 57 months
  Time to Deterioration (TTD) is defined as the time from randomization to first onset of a ≥10-point increase in cough, chest pain, or dyspnea, confirmed by a second adjacent ≥10-point increase from randomization in the same symptom, or confirmed by death within 21 days of a ≥10-point increase from randomization, assessed the European Organization for Research and Treatment of Cancer Lung cancer module (EORTC-QLQ-LC13).
Number of Participants With Treatment-emergent Adverse Events (TEAE) in Participants With Advanced or Metastatic Non Small Cell Lung Cancer (NSCLC) | Up to 57 months
  A TEAE is defined as an AE with a start or worsening date on or after the start date of study treatment until 37 days after the end date of study treatment.
Proportion of Participants Who Are Anti-Drug Antibody (ADA)-Positive (Baseline and Post-Baseline) and Proportion of Participants Who Have Treatment-emergent ADA | Baseline and up to 57 months
  The immunogenicity of Dato-DXd in combination with pembrolizumab will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (254):
- United States (36):
  - Southern Cancer Center Pc, Daphne, Alabama
  - Ironwood Cancer and Research Centers, Chandler, Arizona
  - Arizona Oncology Associates, Pc - Nahoa, Prescott Valley, Arizona
  - Hoag Memorial Hospital Prebyterian, Newport Beach, California
  - Compassionate Cancer Care Medical Group, Riverside, California
  - Sansum Clinic, Santa Barbara, California
  - Ronald Reagan UCLA Medical Center, Santa Monica, California
  - UCHealth Memorial Hospital, Colorado Springs, Colorado
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - Cancer Specialist of North Florida, Jacksonville, Florida
  - Cancer Care Centers of Brevard, Inc., Palm Bay, Florida
  - Woodlands Medical Specialists, Pa, Pensacola, Florida
  - Florida Cancer Specialists-North, St. Petersburg, Florida
  - Emory University - Winship Cancer Institute Wci, Atlanta, Georgia
  - Illinois Cancer Specialists, Niles, Illinois
  - American Oncology Partners of Maryland, Bethesda, Maryland
  - Maryland Oncology Heamtology P.A., Columbia, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute; Inv Drg Svc Pharm, Boston, Massachusetts
  - Dana Farber Cancer Institute At St. Elizabeth'S Medical Center, Brighton, Massachusetts
  - Dana Farber Brigham Cancer Center, Foxborough, Massachusetts
  - Dana Farber At Milford Regional Cancer Center, Milford, Massachusetts
  - Dana Farber/Bwcc in Affiliation With South Shore Hospital, South Weymouth, Massachusetts
  - Astera Cancer Care, East Brunswick, New Jersey
  - Regional Cancer Care Associates LLC, Hackensack, New Jersey
  - North Shore Hematology Oncology Associates dba NY Cancer and Blood Specialists- New Hyde Park, New Hyde Park, New York
  - North Shore Hematology Oncology Associates, Patchogue, New York
  - North Shore Hematology Oncology Associates DBA NY Cancer and Blood Specialists, Port Jefferson Station, New York
  - North Shore Hematology Oncology Associates dba NY Cancer and Blood Specialists - Bronx, The Bronx, New York
  - Texas Oncology, P.A., McAllen, Texas
  - Ut Health San Antonio, San Antonio, Texas
  - Texas Oncology, P.A., Sugar Land, Texas
  - Texas Oncology-Tyler, Tyler, Texas
  - Utah Cancer Specialists IHO Corp, Salt Lake City, Utah
  - Providence Regional Cancer System, Lacey, Washington
  - VA Puget Sound Health Care System, Seattle, Washington
- Argentina (10):
  - Centro de Investigaciones Medicas y Desarrollo LC SRL, Buenos Aires
  - Instituto Alexander Fleming, Buenos Aires
  - Fundacion CENIT para la investigacion en Neurociencias, Ciudad Autonoma de Buenos Aire
  - Hospital de La Comunidad, Mar del Plata
  - Centro de Investigacion Pergamino Sa, Pergamino
  - Instituto de Oncologia de Rosario, Rosario
  - Sanatorio Parque, Rosario
  - Sanatorio Britanico, Rosario
  - Centro Polivalente de Asistencia E Investigacion Clinica Cer San Juan, San Juan
  - Centro de Investigaciones Clinicas. Clinica Viedma S.A., Viedma
- Australia (6):
  - CRSA/ St Andrews Hospital, Adelaide
  - Flinders Medical Centre (Fmc), Bedford Park
  - PSEHOG (Peninsula and South Eastern Haematology and Oncology Group), Frankston
  - St George Public Hospital, Kogarah
  - Southern Medical Day Care Centre, Wollongong
  - Princess Alexandra Hospital, Woolloongabba
- Austria (3):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Klinikum Klagenfurt Pulmologie, Klagenfurt
  - Karl Landsteiner Institut Fã¼R Lungenforschung Und Pneumologische Onkologie C/O Klinik Floridsdorf, Vienna
- Belgium (5):
  - Az Maria Middelares - Campus Maria Middelares, Ghent
  - Centre hospitalier Jolimont-Lobbes, Haine-Saint-Paul
  - Jessa Hospital, Hasselt
  - Cliniques Saint Pierre Ottignies (CSPO), Ottignies
  - Az Nikolaas, Sint-Niklaas
- Brazil (11):
  - Personal Oncologia de Precisao - Cenantron, Belo Horizonte
  - Fundaco Universidade de Caxias Do Sul- Instituto de Pesquisas Em Saude Ips-Ucs, Caxias do Sul
  - Hospital Erasto Gaertner, Curitiba
  - Oncosite - Centro de Pesquisa Clinica Em Oncologia Ltda, Ijuí
  - Clínica de Neoplasias Litoral Ltda, ItajaĂ-
  - Clnica Lacks, Pelotas
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Instituto Nacional de Căncer - Inca, Rio de Janeiro
  - Centro de Estudos E Pesquisa de Hematologia E Oncologia - Cepho, Santo André
  - Instituto de Ensino E Pesquisa Sao Lucas, São Paulo
  - Instituto Do Cancer Brasil - Unidade Taubate, Taubaté
- CHU de Quebec -Universite Laval Hopital de L'Enfant-Jesus, Québec, Canada
- Chile (6):
  - ONCOVIDA, Santiago
  - Centro de Estudios Clinicos Saga Spa, Santiago
  - Orlandi Oncologia, Santiago
  - Fundacion Arturo Lopez Perez, Santiago
  - Centro de Investigaciones Clinicas Vina Del Mar, ViĂąa Del Mar
  - Oncocentro Apys, Viña del Mar
- China (29):
  - Peking University Peoples Hospital, Beijing
  - Peking University Cancer Hospital Beijing Cancer Hospital Beijing Institute For Cancer Research, Beijing Sheng
  - Cangzhou Peoples Hospital, Cangzhou
  - First Affiliated Hospital of Medical College of Jilin University, Changchun
  - Jilin Cancer Hospital, Changchun
  - Hunan Cancer Hospital, Changsha
  - University of Electronic Science Technology of China UESTC - Sichuan Cancer Hospital Institute SIC, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - Fujian Medical University - Union Hospital Foochow Christian Union Hospital, Fuzhou
  - The First Affiliated Hospital Sun Yat-Sen University, Guangzhou
  - Affiliated Cancer Hospital and Insititute of Guangzhou Medical University, Guangzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou
  - The First Affiliated Hospital of College of Medicine Zhejiang University, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - An Hui Cancer Hospital, Hefei
  - Inner Mongolia Medical University- the Affiliated Hospital, Hohhot
  - Jiamusi Cancer Hospital, Jiamusi
  - Linyi Cancer Hospital, Linyi
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Zhongda Hospital, Southeast University, Nanjing
  - Shanghai Chest Hospital, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Liaoning Cancer Hospital & Institute, Shenyang
  - The First Affiliated Hosptial of Xinjiang Medical University, Ürümqi
  - Union Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - The First Affiliate Hospital of Xi'An Jiaotong University, Xi'an
  - Xiangyang Central Hospital, Xianyang
  - Henan Cancer Hospital, Zhengzhou
- Czechia (2):
  - FN Brno Klinika Nemoci Plicnich a TBC, Brno
  - Fakultni nemocnice Olomouc FNOL, Olomouc
- France (15):
  - Sainte-Catherine Institut du Cancer Avignon-Provence, Avignon
  - Hopital Jean Minjoz - CHU de Besancon, Besançon
  - Chu de Bordeaux - Hopital Saint Andre, Bordeaux
  - Centre Hospitalier Universitaire, CHU, de Poitiers, France
  - Hopital Lyon Sud, Lyon
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Aphm - Hopital Nord, Marseille
  - Chu de Montpellier, Montpellier
  - Chu de Nantes, Nantes
  - Hopital Prive Du Confluent, Nantes
  - Institut Curie, Paris
  - Tenon Hospital, Paris
  - CHU de Rennes - Hopital Pontchaillou, Rennes
  - Hôpital Foch, Suresnes
- Germany (9):
  - Evangelische Lungenklinik Berlin, Berlin
  - Klinikum Chemnitz, Chemnitz
  - Universitaetsklinikum Essen, Essen
  - Klinikum Esslingen Gmbh, Esslingen am Neckar
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - University Hospital Giessen, ZIM IV, Giessen
  - External pharmacy Fortuna Herstellung GmbH of main site Universitaetsmedizin Mannheim, Mannheim
  - Ludwig-Maximilians University Hospital of Munich, Munich
  - University Hospital Mănster, Münster
- Greece (9):
  - Sotiria General Hospital of Chest Diseases, Athens
  - Metropolitan Hospital - Athens, Athens
  - University General Hospital of Heraklion, Heraklion
  - University Hospital of Ioannina Uhi, Ioannina
  - Metropolitan Hospital, Neo Faliro
  - Olympion Hospital, Pátrai
  - Euromedica General Clinic of Thessaloniki, Thessaloniki
  - St. Luke's Hospital, Thessaloniki
  - Bioclinic Thessaloniki (Galinos Clinic), Thessalonki
- Hong Kong (3):
  - Tuen Mun Hospital, Hong Kong
  - Prince of Wales Hospital / The Chinese University of Hong Kong, Hong Kong
  - Queen Mary Hospital, Pok Fu Lam
- Hungary (6):
  - National Koranyi Institute For Pulmonology, Budapest
  - Veszprem Megyei Tudogyogyintezet Farkasgyepu, Farkasgyepű
  - Bkmk Hospital, KecskemĂŠt
  - Fejer Megyei Szent Gyorgy Korhaz Pulmonologiai Osztaly, Székesfehérvár
  - Hetenyi G Korhaz, Onkologiai Kozpont, Szolnok
  - Reformatus Pulmonologiai Centrum, Törökbálint
- Italy (7):
  - Istituto Di Candiolo Irccs, Candiolo
  - Ospedale San Luca, Lucca
  - Azienda Ospedaliero - Universitaria San Luigi Gonzaga, Orbassano
  - IFO Regina Elena, Rome
  - Ospedale S. Maria Della Misericordia, Udine
  - Asst Sette Laghi, Varese
  - Azienda Ospedaliera Universitaria Integrata Verona Ospedale Borgo Roma Crc - Centro Ricerche Clinich, Verona
- Japan (26):
  - NHO Shikoku Cancer Center, Ehime
  - Kurume University Hospital, Fukoka
  - Kyushu Cancer Center, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Teine Keijinkai Hospital, Hokkaido
  - Hyogo Medical University Hospital, Hyōgo
  - Kanazawa University Hospital, Ishikawa
  - Kanagawa Cancer Center, Kanagawa
  - Kitasato University hospital, Kanagawa
  - Social Welfare Organization Saiseikai Imperial Gift Foundation, Inc. Saiseikai Kumamoto Hospital, Kumamoto
  - University Hospital Kyoto Prefectual University of Medicine, Kyoto
  - Matsusaka Municipal Hospital, Mie
  - Sendai Kousei Hospital, Miyagi
  - Niigata Cancer Center Hospital, Niigata
  - Osaka International Cancer Institute, Osaka
  - Osaka Toneyama Medical Center, Osaka
  - Kansai Medical University Hospital, Osaka
  - NHO Kinki-Chuo Chest Medical Center, Osaka
  - Dokkyo Medical University Hospital, Tochigi
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Tokyo
  - Juntendo University Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Toho University Omori Medical Center, Tokyo
  - Iwakuni Clinical Center, Yamaguchi
  - Yamaguchi-Ube Medical Center, Yamaguchi
  - Yamanashi Prefectural Central Hospital, Yamanashi
- Mexico (5):
  - Cryptex Investigacion Clinica Sa de Cv, Cuauhtémoc
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara
  - Health Pharma Professional Research S.A de C.V., Mexico City
  - Instituto Nacional de Cancerologia, Mexico City
  - Centro de Investigacion Clinica de Oaxaca CICLO, Oaxaca City
- Netherlands (3):
  - Jeroen Bosch Ziekenhuis Jbz, 's-Hertogenbosch
  - Amphia Ziekenhuis, Breda
  - Leiden University Medical Center, Leiden
- Poland (6):
  - II Klinika Chorob Pluc i Gruzlicy, Bialystok
  - Centrum Terapii Wspolczesnej, Lodz
  - Instytut Centrum Zdrowia Matki Polki (Iczmp), Lodz
  - SPSK4, Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie, Lublin
  - Med Polonia Sp. Z O.O., Poznan
  - Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw
- Portugal (3):
  - Fundacao Champalimaud, Lisbon
  - IPO Porto Francisco Gentil, E.P.E., Porto
  - Hospital CUF Porto, Porto
- Romania (5):
  - Institute of Oncology Prof. Dr. Ion Chiricuta, Cluj-Napoca
  - Onco Clinic Consult Sa, Craiova
  - Centrul de Oncologie Sfantu Nectarie, Craiova
  - SC Oncomed SRL, Jud Timis
  - Oncocenter Oncologie Clinica S.R.L, Timișoara
- South Korea (9):
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National University Chilgok Hospital, Daegu
  - Samsung Medical Center, Gangnam-Gu
  - National Cancer Center, Goyang-si
  - Gyeongsang National University Hospital, Jinju-si Gyeongsangnam-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Yonsei University Health System - Severance Hospital, Seoul
  - The Catholic Univ. of Korea, Seoul St. Marys Hospital, Seoul
- Spain (12):
  - Vall Hebron University Hospital, Barcelona
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Hospital Universitario Arnau de Vilanova, Lleida
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Regional Universitario Malaga, Málaga
  - CHUO, Ourense
  - Hosp Univ Virgen Macarena, Seville
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Universitario y Politecnico de La Fe, Valenica
  - Hospital Universitario Miguel Servet, Zaragoza
- Switzerland (3):
  - Kantonsspital Baselland, Liestal
  - Kantonsspital St. Gallen, Sankt Gallen
  - Spital Sts Ag, Thun
- Taiwan (9):
  - Changhua Christian Hospital, Changhua
  - China Medical University Hospital, Hsia
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Thailand (6):
  - Faculty of Medicine Chulalongkorn University, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Chiang Mai University CMU - Maharaj Nakhon Chiang Mai Hospital Nakorn Chiang Mai Hospital, Chiang Mai
  - Prince of Songkla University PSU - Faculty of Medicine, Hat Yai
  - Khon Kaen University - Faculty of Medicine-Srinagarind Hospital, Nonthaburi
- Turkey (Türkiye) (8):
  - Baskent University, Adana
  - Ankara Bilkent City Hospital, Ankara
  - Akdeniz University Hospital, Antalya
  - Medipol Mega University Hospital, Bağcılar
  - Ege Universitesi Gogus Hastaliklari Poliklinigi, Bornova-Izmir
  - Memorial Ankara Hospital, Cankaya/Ankara
  - Istanbul Medeniyet University Medical Faculty, Istanbul
  - Adana Acibadem Hospital, Seyhan
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Okamoto I, Kuyama S, Girard N, Lu S, Franke F, Li Z, Danchaivijitr P, Han JY, Sun JM, Sugawara S, Pan E, Ren N, Chen A, Rajagopalan R, Lisberg AE. TROPION-Lung07: Phase III study of Dato-DXd + pembrolizumab +/- platinum-based chemotherapy as 1L therapy for advanced non-small-cell lung cancer. Future Oncol. 2024;20(37):2927-2936. doi: 10.1080/14796694.2024.2409621. Epub 2024 Oct 29. PMID 39469838